CLINICAL TRIAL: NCT04792866
Title: 3D FLAIR Versus Coronal T2-WI MRI in Detecting Optic Neuritis in Patients Presenting With Acute Visual Loss and Otherwise Normal Ophthalmological Examination
Brief Title: 3D FLAIR Versus Coronal T2-WI MRI in Detecting Optic Neuritis (FLACON)
Acronym: FLACON
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: CE_20200204_1_ALR
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Optic Neuritis; Multiple Sclerosis; Encephalopathy
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis; Brain Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Comparing 3D FLAIR versus Coronal T2-WI MRI in detecting Optic Neuritis

SUMMARY:
3D FLAIR, 3D T1 FAT SAT, coronal T2 and coronal T1 dixon sequences were usually used to assess visual deficits in MRI. Optic nerve examination is preferably performed using a coronal T2 sequence in order to detect a hypersignal suggestive of inflammation whereas brain examination is preferably performed using a 3D FLAIR sequence to highlight signs of spatial dissemination and lesions suggestive of multiple slerosis (MS).

Recently, a study based on a small number of patients showed the interest of 3D FLAIR in the detection of the hypersignal of the optic nerve.The objective of this retrospective study is to determine whether a single 3D FLAIR sequence allows simultaneous exploration of the optic nerve and the brain for the positive diagnosis of optic neuropathy and/or MS.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Decrease in visual acuity explored in MRI between january 2018 and january 2020

Exclusion Criteria:

* Past history of episode of Optic neuritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute visual loss and explored by MRI
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Detection of optic neuropathies using MRI | 1 hour
  MRI comparison of the diagnostic performance of the 3D FLAIR sequence and the T2 coronal in the detection of optic neuropathies.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Île-de-France Region, France